CLINICAL TRIAL: NCT00005078
Title: Phase I Dose Escalation Study of Tirapazamine (NSC 130181) in Combination With Carboplatin and Paclitaxel in Advanced Malignant Solid Tumors
Brief Title: Tirapazamine, Carboplatin, and Paclitaxel in Treating Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 99139; U01CA062505 (NIH); P30CA033572 (NIH); CHNMC-PHI-22; CHNMC-IRB-99139; NCI-T99-0068; CDR0000067685 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-04-06; First posted 2003-05-16 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Carboplatin; Paclitaxel; Tirapazamine

INTERVENTIONS:
Drug: carboplatin
Drug: paclitaxel
Drug: tirapazamine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining tirapazamine, carboplatin, and paclitaxel in treating patients who have advanced malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of tirapazamine in combination with carboplatin and paclitaxel in patients with advanced solid tumors who have or have not received prior chemotherapy.
* Assess the toxicity and preliminary efficacy of this regimen in these patients.
* Determine the pharmacokinetic profile of this regimen in these patients.
* Investigate potential predictors of response by studying patient tissue specimens after receiving this regimen.

OUTLINE: This is a dose-escalation study of tirapazamine. Patients are stratified according to prior chemotherapy status (previously untreated vs previously treated).

Patients receive tirapazamine IV over 2 hours, paclitaxel IV over 3 hours, and carboplatin IV over 30 minutes. Treatment continues every 21 days for a maximum of 8 courses in the absence of unacceptable toxicity or disease progression. Some patients may continue therapy in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tirapazamine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients in the previously untreated stratum are treated at the MTD.

Patients are followed indefinitely.

PROJECTED ACCRUAL: A total of 36-68 patients (18-34 per stratum) will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced or metastatic malignant solid tumor not curable by resection or other standard therapy
* No symptomatic brain metastases

  * Brain metastases allowed provided controlled with surgical excision and/or radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm3
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal

Renal:

* Creatinine normal
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV congestive heart failure

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No history of allergic reactions to appropriate diuretics or antiemetics administered in conjunction with protocol chemotherapy (e.g., 5-HT3 antagonists)
* No other concurrent uncontrolled illness that would preclude study therapy
* No medical, social, or psychological factors that would preclude study therapy
* No clinically significant hearing loss

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas) and recovered
* No more than 2 prior chemotherapy regimens
* No prior combination paclitaxel and carboplatin

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* At least 30 days since other prior investigational drugs
* No other concurrent anticancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Shibata, MD, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California

REFERENCES:
- [Result] Lara PN Jr, Frankel P, Mack PC, Gumerlock PH, Galvin I, Martel CL, Longmate J, Doroshow JH, Lenz HJ, Lau DH, Gandara DR. Tirapazamine plus carboplatin and paclitaxel in advanced malignant solid tumors: a california cancer consortium phase I and molecular correlative study. Clin Cancer Res. 2003 Oct 1;9(12):4356-62. PMID 14555506